CLINICAL TRIAL: NCT01774591
Title: Effect of Azilsartan on Aldosterone in Postmenopausal Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-1179
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Post Menopause; Female; Obese
MeSH Terms: conditions — Hypertension; Obesity | interventions — azilsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- azilsartan medoximil. (Active Comparator): Subjects randomized to azilsartan medoximil arm will take 80 mg of azilsartan medoximil tablets by mouth each day.
  Interventions: Drug: Azilsartan medoximil
- Placebo (Placebo Comparator): Subjects randomized to the placebo arm will take 80 mg of placebo tablets by mouth each day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan medoximil — All subjects were randomized to 80mg azilsartan medoxomil (azilsartan) daily or placebo and followed for six months.
  Other Names: Edarbi
  Arms: azilsartan medoximil.
Drug: Placebo — All subjects were randomized to 80mg azilsartan medoxomil (azilsartan) daily or placebo and followed for six months.
  Arms: Placebo

SUMMARY:
The purpose of the research is to evaluate the effect of azilsartan medoximil on blood pressure and urinary aldosterone levels in postmenopausal females.

DETAILED DESCRIPTION:
The study is a randomized, placebo-controlled trial of post-menopausal females with stage 1 hypertension. The goal is to randomize 40 post-menopausal females with stage 1 hypertension and assess whether azilsartan reduces urinary aldosterone levels. We will compare subjects having azilsartan medoximil (treatment group) with placebo group. Additionally, a small sub-study comparing pre-menopausal and post-menopausal female aldosterone levels was performed as well as the presence of aldosterone production in fat cell cultures of a subset of 3 patients in the randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 45-70
* Post-menopause: have not had a menstrual period for one year or more
* Diagnosed with Stage 1 hypertension
* Body Mass Index (BMI) greater than or equal to 28

Exclusion Criteria:

* Male
* Diagnosed with Stage 2 hypertension
* Stage 1 hypertension requiring more than one agent
* Pregnancy or attempting pregnancy
* Use of oral contraceptive pills
* Use of hormone replacement therapy
* Use of steroids
* Stage 3 or greater kidney disease
* Diabetes mellitus
* untreated hypothyroidism or hyperthyroidism
* primary hyperaldosteronism
* Cushing's disease
* obstructive sleep apnea
* chronic illness, e.g. chronic liver disease
* NYHA class III or greater heart failure
* moderate to severe lung disease

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Bakris, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Azilsartan Medoximil.: Subjects randomized to azilsartan medoximil arm will take 80 mg of azilsartan medoximil tablets by mouth each day and followed for six months.
- Placebo: Subjects randomized to the placebo arm took 80 mg of placebo tablets by mouth each day and followed for six months.
Period: Overall Study
Arm/Group | Azilsartan Medoximil. | Placebo
Started | 10 | 11
Completed | 9 | 7
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoximil. | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [56 to 63] | 55 [53 to 57] | 57 [54 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 24-hour BP (Systolic)
Description: To evaluate the effect of an angiotensin receptor blocker (azilsartan medoximil) on blood pressure in postmenopausal females.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoximil. | Placebo
Number analyzed (Participants) | 10 | 11
mmHg | 113 (14) | 129 (904)

2. Secondary Outcome: Difference in 24-hour Urine Aldosterone Change From Baseline
Description: To evaluate the effect of an angiotensin receptor blocker (azilsartan medoximil) on urinary aldosterone levels in postmenopausal females
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage of changes
Arm/Group | Azilsartan Medoximil. | Placebo
Number analyzed (Participants) | 10 | 11
percentage of changes | -47.3 (32.9) | -5.3 (52.3)

3. Primary Outcome: 24-hour BP (Diastolic)
Description: as for outcome 1
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoximil. | Placebo
Number analyzed (Participants) | 10 | 11
mmHg | 75 (8.8) | 89 (11)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Azilsartan Medoximil. | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 3/10 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoximil. (N=10) | Placebo (N=11)
Hypotension (Vascular disorders) | 1 | 0
Edema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No